CLINICAL TRIAL: NCT00670605
Title: VICC Adolescent and Young Adult Oncology Review
Brief Title: Cancer Occurrence and Outcome in Young Patients Undergoing Cancer Treatment at the Vanderbilt-Ingram Cancer Center
Status: Terminated | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000584244; P30CA068485 (NIH); VU-VICC-PED-0732; VU-VICC-070568
Record Dates: First submitted 2008-05-01; First posted 2008-05-02 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2011-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; unspecified childhood solid tumor, protocol specific

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: medical chart review
Other: study of socioeconomic and demographic variables

SUMMARY:
RATIONALE: Gathering information about the number of young patients with cancer and the outcome of these patients may help doctors learn more about cancer.

PURPOSE: This research study is looking at the medical records of young patients undergoing cancer treatment at the Vanderbilt-Ingram Cancer Center to determine how often cancer occurs and the outcome of these patients.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the number of patients between 15 and 30 years old who are treated for newly diagnosed cancer at the Vanderbilt-Ingram Cancer Center (VICC), in middle Tennessee, and in the state of Tennessee between 1990 and 2005.
* To determine the outcomes of these patients.
* To determine the number of these patients enrolled on clinical trials at VICC.
* To compare the outcomes of these patients when treated on a trial versus not treated on a trial provided they have the same disease.
* To compare the number of these patients who are treated on a clinical trial when they are first seen at Vanderbilt Children's Hospital vs Vanderbilt University Hospital.
* To determine referral patterns of these patients to VICC.
* To compare the outcomes of these patients who are treated at VICC vs middle Tennessee vs the state of Tennessee vs the entire nation.
* To determine the reason for not enrolling on a clinical trial.

OUTLINE: Cancer cases taken from the Vanderbilt-Ingram Cancer Center (VICC) Registry and the Tennessee Cancer Registry are examined for number and types of cancer, mortality rates broken down by county and health department region, electronic medical records, and treatment outcomes. Data is analyzed for comparison of number of new cancer patients, mortality rates, and referral patterns at VICC versus number of new cancer patients in the region, state, and country.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cancer

  * Newly diagnosed disease from 1990 to 2005
  * 15 to 30 years old at the time of cancer diagnosis
* Must live in the state of Tennessee

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Newly diagnosed
Sampling Method: Probability Sample
Dates: Start 2007-06; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with newly diagnosed cancer from 1990 to 2005 and treated at Vanderbilt-Ingram Cancer Center (VICC), in middle Tennessee, and the state of Tennessee
Comparison of outcomes
Number of patients enrolled in clinical trials at VICC
Outcomes of patients treated on a trial vs those not treated with the same disease
Comparison of number of patients treated at Vanderbilt Children's Hospital vs Vanderbilt University Hospital
Referral patterns
Reason for not enrolling on a clinical trial

CONTACTS AND LOCATIONS:
Overall Officials: Anderson B. Collier, MD, Study Chair — Vanderbilt Children's Hospital
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee